CLINICAL TRIAL: NCT06476184
Title: A Pragmatic Randomized Phase III Trial to Assess the Utility of Adjusting Chemotherapy Dose & Dosing Schedule With the SALVage Weekly Dose-dense Regimen in Patients With Poor Prognostic OVARian Cancers Based on the Tumor Unfavorable Primary Chemosensitivity and Incomplete Debulking Surgery
Brief Title: Utility of Adjusting Chemotherapy Dose & Dosing Schedule With the SALVage Weekly Dose-dense Regimen in Patients With Poor Prognostic OVARian Cancers Based on the Tumor Unfavorable Primary Chemosensitivity and Incomplete Debulking Surgery
Acronym: SALVOVAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Collaborators: Horizon 2020 - European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-508260-30-01; RECF-005636 (Other: INCA)
Record Dates: First submitted 2024-06-05; First posted 2024-06-26 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer
Keywords: chemotherapy; poor prognostic; unfavorable primary chemosensitivity; incomplete debulking surgery; KELIM
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Patients will be randomized 1:1:
  * Experimental arm: Densification of the chemotherapy administration dose and dosing schedule of carboplatin-paclitaxel (carboplatin AUC 5 every 3 weeks on day 1 and paclitaxel 80 mg/m2 every week, on day 1, day 8, and day 15, with 3 week-cycles) for 3 cycles
    +/- combined with daily sub-cutaneous administrations of GCSF (Granulocyte Colony-Stimulating Factor) 30 MUI days 3 to 5, & 10 to 12, & 17 to 19 (at investigator discretion, as per standard of care)
  * Standard arm: Continuation of the same 3-weekly carboplatin-paclitaxel, as administered during the neo-adjuvant chemotherapy +/- combined with peg-GCSF or GCSF daily sub-cutaneous administrations, at investigator discretion, as per standard of care.
  Of note, bevacizumab addition in both arms is required in countries where it is available as per standard of care, according to country health coverage policy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental): Densification of the chemotherapy administration dose and dosing schedule of carboplatin-paclitaxel (carboplatin AUC 5 every 3 weeks on day 1 and paclitaxel 80 mg/m2 every week, on day 1, day 8, and day 15, with 3 week-cycles) for 3 cycles
  +/- combined with daily sub-cutaneous administrations of GCSF 30 MUI days 3 to 5, & 10 to 12, & 17 to 19 (at investigator discretion, as per standard of care).
  Interventions: Drug: Carboplatin; Drug: Paclitaxel
- Standard (Active Comparator): Continuation of the same 3-weekly carboplatin-paclitaxel, as administered during the neo-adjuvant chemotherapy
  +/- combined with peg-GCSF or GCSF daily sub-cutaneous administrations, at investigator discretion, as per standard of care.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Carboplatin — Patients will be randomized 1:1:
  * Experimental arm: Densification of the chemotherapy administration dose and dosing schedule of carboplatin-paclitaxel (carboplatin AUC 5 every 3 weeks on day 1 and paclitaxel 80 mg/m2 every week, on day 1, day 8, and day 15, with 3 week-cycles) for 3 cycles
  * Standard arm: Continuation of the same 3-weekly carboplatin-paclitaxel, as administered during the neo-adjuvant chemotherapy
Drug: Paclitaxel — Patients will be randomized 1:1:
  * Experimental arm: Densification of the chemotherapy administration dose and dosing schedule of carboplatin-paclitaxel (carboplatin AUC 5 every 3 weeks on day 1 and paclitaxel 80 mg/m2 every week, on day 1, day 8, and day 15, with 3 week-cycles) for 3 cycles
  * Standard arm: Continuation of the same 3-weekly carboplatin-paclitaxel, as administered during the neo-adjuvant chemotherapy

SUMMARY:
SALVOVAR will be a pragmatic open-label multicenter randomized phase III trial (ratio 1:1) comparing the efficacy of the salvage weekly dose-dense regimen with those of the continuation of the standard regimen.

DETAILED DESCRIPTION:
SALVOVAR is a pragmatic open-label multicenter randomized phase III trial (ratio 1:1) comparing the efficacy of the salvage weekly dose-dense regimen with those of the continuation of the same standard regimen as given during neo-adjuvant period. The randomization will be stratified on the main clinical prognostic factors assumed to impact the efficacy of the assessed arms and the overall survival:

1. Bevacizumab: planned administration: Yes, vs No
2. BRCA mutation: planned administration: Yes, vs No/Unknown
3. KELIMTM strate within unfavorable KELIM subgroup: very unfavorable < 0.7, vs moderately unfavorable [0.7-1.0[

The trial will be pragmatic, as it aims at confirming the superiority of the adjusted chemotherapy compared to the continuation of the standard chemotherapy in routine clinical practice, in a population of ovarian cancer patients close to the real-life clinical activity with few selection criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed high-grade epithelial (serous, endometrioid, or carcinosarcoma with a ≥30% epithelial tumor component) ovarian, primary peritoneal, or fallopian-tube carcinoma
2. Adult patient aged ≥ 18 years old
3. Advanced stage III or IV disease
4. Treated with 3 to 4 neo-adjuvant cycles of standard 3-weekly carboplatin-paclitaxel regimen in first-line setting, and characterized by:

   * Unfavorable standardized KELIMTM score < 1.0 calculated with the KELIMTM academic tool and available for free on internet site (https://www.biomarker-kinetics.org/CA-125-neo) (poor primary chemosensitivity)
   * Not amenable to complete interval debulking surgery (incomplete interval debulking surgery attempt, or disease not operated at all because considered not amenable to complete surgery by surgeon) Of note, a pre-screening inclusion before the start of neo-adjuvant chemotherapy is encouraged as a way of prospectively assessing the CA-125 longitudinal kinetics and surgery evaluation, and subsequently selecting the patients for the randomization sequence
5. ECOG performance status 0 or 1 (see appendix 2)
6. Adequate organ and bone marrow function for weekly-dense chemotherapy: red blood cells (baseline Hemoglobin ≥8 g/dL without red blood cell transfusion within 3 weeks before the blood work), white blood cells (Absolute neutrophil count (ANC) ≥1500 cells/mm3) and platelets (Platelet count ≥100,000/mm3),
7. Adequate renal and liver functions

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × upper limit of normal (ULN), or ≤5 × ULN in context of liver metastases
   * Total bilirubin ≤1.5 × ULN (patients with Gilbert's are eligible if total bilirubin ≤3 × ULN)
   * Albumin ≥3 g/dL
   * Creatinine clearance ≥40 mL/min/1.73 m2 (measured or estimated, ideally with CKD-EPI formula on https://www.kidney.org/professionals/kdoqi/gfr_calculator)
8. Patients who gave its written informed consent to participate to the study
9. Patients affiliated to a social insurance regime
10. Patients willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up

Exclusion Criteria:

1. Low-grade endometrioid, clear cell, mucinous, or sarcomatous histology, or mixed tumors containing any of these histologies, or low-grade or borderline ovarian tumor. Contraindication to the drugs assessed in the SALVOVAR trial (carboplatin, paclitaxel, GCSF)
2. Previous treatment with bevacizumab during initial standard neo-adjuvant chemotherapy
3. Has primary platinum-refractory disease, defined as disease that has progressed during the neo-adjuvant chemotherapy
4. Patients with concomitant cancer, except: adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥ 5 years
5. Treatment with other investigational agents in clinical trials.
6. Clinically significant uncontrolled condition(s) which, in the opinion of the Investigator, may confound the results of the trial or interfere with the patient's safety or participation, including but not limited to:

   * Unstable angina.
   * Myocardial infarction within 6 months of first dose.
   * Uncontrolled and/or severe concomitant diseases (uncontrolled hypertension, ≥ Grade 3 (per CTCAE v5.0) arrhythmia, heart failure, cirrhosis).
   * Active infectious disease requiring IV therapy (bacteria, viruses) within 2 weeks of first dose.
   * Gastric-outlet obstruction.
   * Small bowel obstruction (SBO) defined as computed tomography (CT) scan showing: Dilated loops of small bowel ≤12 weeks of study entry, symptomatic ascites/effusions requiring paracentesis or thoracentesis ≤30 days of study entry.
7. Known psychiatric disorder that would interfere with trial compliance.
8. Pregnant or lactating patients or patients expecting to conceive children within the projected duration of the trial.
9. Patient deprived of liberty, under guardianship, or under curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients operated with late complete debulking surgery | From the date of randomization until patients operated with late complete debulking surgery, assessed up 100 days
  To demonstrate the superiority in terms of efficacy of a densification of the chemotherapy with the salvage weekly dose-dense carboplatin-paclitaxel regimen compared to the continuation of the standard 3-weekly carboplatin-paclitaxel, in ovarian cancer patients found to have a poor prognostic disease (characterized by a poor chemosensitivity, with an unfavorable KELIMTM score < 1.0, and a disease not amenable to complete interval debulking surgery) after 3 cycles of standard neo-adjuvant chemotherapy.
Overall survival (OS) | From the date of randomization until death due to any cause, assessed up to 5 years
  To demonstrate the superiority in terms of efficacy of a densification of the chemotherapy with the salvage weekly dose-dense carboplatin-paclitaxel regimen compared to the continuation of the standard 3-weekly carboplatin-paclitaxel, in ovarian cancer patients found to have a poor prognostic disease (characterized by a poor chemosensitivity, with an unfavorable KELIMTM score < 1.0, and a disease not amenable to complete interval debulking surgery) after 3 cycles of standard neo-adjuvant chemotherapy.

SECONDARY OUTCOMES:
Percentage of patients operated with late complete debulking surgery, regardless of the number of chemotherapy cycles received | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To compare the efficacy, in term of percentage of patients operated with late complete debulking surgery, between the salvage weekly dose-dense regimen and the standard regimen, regardless of the number of chemotherapy cycles received.
Overall response rate according to RECIST V1.1 in the whole population | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To compare the efficacy of the salvage weekly dose-dense regimen with those of the standard regimen in terms of:
  * Radiological response after 3 cycles of treatment, based on the best radiological response using RECIST criteria
  * Progression-free survival
Progression-free survival in the whole population | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To compare the efficacy of the salvage weekly dose-dense regimen with those of the standard regimen in terms of:
  • Radiological response after 3 cycles of treatment, based on the best radiological response using RECIST criteria
Percentage of patients treated with a subsequent maintenance treatment with a PARP inhibitor (%) in the whole population | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To assess the impact of the adjustment to the salvage weekly dose-dense regimen on the rate of subsequent prescription of PARP inhibitors (since these drugs are indicated in patients with complete or partial response to platinum-based chemotherapy) in terms of survival.
Progression-free survival and overall survival in these patients compared to those not treated with PARP inhibitor | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To assess the impact of the adjustment to the salvage weekly dose-dense regimen on the rate of subsequent prescription of PARP inhibitors (since these drugs are indicated in patients with complete or partial response to platinum-based chemotherapy) in terms of survival.
To assess the impact of adding bevacizumab to chemotherapy (salvage or standard arm) on the efficacy outcomes In the population of patients treated with bevacizumab: - Overall response rate according to RECIST V1.1 | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To assess the impact of adding bevacizumab to chemotherapy (salvage or standard arm) on the efficacy outcomes
Adverse events graded according to the NCI Common Terminology Criteria Adverse Event Version 5.0 | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To compare the safety profiles of the salvage weekly dose-dense chemotherapy arm with those of the standard 3-weekly carboplatin-paclitaxel with/without bevacizumab, based on the observed adverse-events
To assess the impact of adding bevacizumab to chemotherapy on the efficacy outcomes In the population of patients treated with bevacizumab: - Progression-free survival & overall survival according to RECIST V1.1 | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To assess the impact of adding bevacizumab to chemotherapy (salvage or standard arm) on the efficacy outcomes
To assess the impact of adding bevacizumab to chemotherapy on the efficacy outcomes In the population of patients treated with bevacizumab: - Percentage of patients operated with a late complete debulking surgery (%) | from the date of randomization until objective tumor progression based on RECIST 1.1, or death due to any cause, whichever occurs first assessed up to 3 years
  To assess the impact of adding bevacizumab to chemotherapy (salvage or standard arm) on the efficacy outcomes

OTHER OUTCOMES:
Quality of life questionnaires | from date of randomization through study completion, an average of 3 years
  To compare the quality of life and patient-reported outcomes of the salvage chemotherapy arm with those of the standard regimen
Perceptions of the patient-doctor relationship in patients offered bevacizumab/debulking surgery/PARPi | From 4-8 weeks after a decision on bevacizumab (approx. at randomization date) through end of follow-up (2-3 years after inclusion, depending on debulking surgery)
  Measure of patient-doctor relationship: The Patient-Doctor Relationship Questionnaire measures patient perceptions of the patient-doctor relationship. Participants rate the level of helpfulness, time, trust, understanding, dedication, agreement, availability, contentment, and accessibility of their healthcare provider. All nine items are rated on a five-point Likert scale from 1 (Not at all appropriate) to 5 (totally appropriate). Mean scores are calculated, and higher scores indicate a better perceived doctor-patient relationship.
Satisfaction with decision-making process in patients offered bevacizumab/debulking surgery/PARPi | From 4-8 weeks after a decision on bevacizumab (approx. at randomization date) through end of follow-up (2-3 years after inclusion, depending on debulking surgery)
  Measure of satisfaction with care: One self-generated item developed on the basis of the literature will ask patients in general how they would rate the care they received for their ovarian cancer treatment during the past three months, using a five-point scale from 1 (poor) to 5 (excellent). A higher score reflects a higher satisfaction with their care.
Satisfaction with decision-making process in patients offered bevacizumab/debulking surgery/PARPi | From 4-8 weeks after a decision on bevacizumab (approx. at randomization date) through end of follow-up (2-3 years after inclusion, depending on debulking surgery)
  Measure of decision satisfaction: The Satisfaction with Decision scale measures a patient's level of satisfaction with healthcare decisions. It consists of six statements to which respondents are asked to indicate their level of agreement using a five-point scale, from 1 (strongly disagree) to 5 (strongly agree). Total scores are summed, with higher scores indicating greater decisional satisfaction.
Emotional wellbeing following the decision-making process in patients offered bevacizumab/debulking surgery/PARPi | From 4-8 weeks after a decision on bevacizumab (approx. at randomization date) through end of follow-up (2-3 years after inclusion, depending on debulking surgery)
  To determine the impact of the decision-making process on emotional wellbeing in the short- and medium-term, among patients who have participated in decision-making regarding bevacizumab as a chemosensitizer, late debulking surgery in the case of favorable response to chemotherapy, or PARP inhibitors and/or bevacizumab as maintenance treatment.
  Measure of emotional wellbeing: Six self-generated items will be used to measure the concept of eudaimonic or hedonic wellbeing. A 10-point scale from 1 (not at all) to 10 (very much so) will gauge perceptions of feeling hopeful, peaceful, grateful, comforted, connected, and content over the past week, presented as single-word descriptors. Mean scores will be calculated for each subscale, and a mean across all items will be derived to reflect overall emotional wellbeing. Higher scores indicate higher levels of emotional wellbeing.
Treatment beliefs in patients offered bevacizumab/PARPi | From 4-8 weeks after a decision on bevacizumab (approx. at randomization date) through end of follow-up (2-3 years after inclusion, depending on debulking surgery)
  Measure of treatment beliefs: For patients prescribed PARP inhibitors and/or bevacizumab, four items will be presented to measure treatment beliefs in relation to these treatments. These items are adapted from a Treatment Beliefs Questionnaire originally developed for patients with low back pain, which has been adapted for the current setting with permission. This self-report scale consists of four items assessing perceptions of credibility, effectiveness, concerns, and individual fit of treatment, which are rated on a five-point scale from (1) strongly disagree to (5) strongly agree. Higher scores for each item indicate more positive beliefs about the treatment (with responses on the 'concerns' item being reverse scored).
Self-reported adherence to PARPi in patients offered PARPi | From 4-8 weeks after a decision on PARPi (approx. at end of chemotherapy) through end of follow-up (2-3 years after inclusion, depending on debulking surgery)
  Measure of treatment (PARPi) adherence: For patients prescribed PARP inhibitors, a three-item scale will be used to measure adherence to PARPi and bevacizumab. Patients will be asked about the number of days in which they missed at least one dose of the treatment (answered numerically), the frequency with which they took their medication in the way they were supposed to over the previous 30 days (rated on a 6-point scale from never to always), and their rating of how 'good a job' they did at taking their medication in the way recommended over the previous 30 days (rated on a 6-point scale from very poor to excellent). Responses will be linearly transformed to a 0-100 scale for analyses, with 0 representing the worst adherence and 100 the best. Summary scores will be calculated as the mean of the three items.
Percentage of patients with BRCA (BReast CAncer) mutation (%) | from date of randomization through study completion, an average of 5 years
  Number of patients with BRCA mutation involved in homologous recombination (%)
Percentage of patients with BRCA wild-type HRD (Homologous Recombination Deficiency) disease (%) | from date of randomization until end of study, for a period of 5 years
  Number of patients with BRCA wild-type HRD mutation involved in homologous recombination (%)
Percentage of patients with BRCA wild-type HRP (Homologous Recombination Proficient) disease (%) | from date of randomization through study completion, an average of 3 years
  Number of patients with BRCA wild-type HRP mutation involved in homologous recombination (%)
Tests/assays used (names, proprietary) | from date of randomization until end of study, through study completion, an average of 3 years
  Name of tests/assays used in real-life setting
Percentage of tests/assays used (names, proprietary) (%) | from date of randomization until end of study, through study completion, an average of 3 years
  Percentage of tests/assays used in real-life setting (%)
Incremental cost-utility ratio | from date of randomization until end of study, for a periof of 5 years
  To assess the cost-utility evaluations of the experimental treatment (medico-economic evaluation) in the French context Salvage weekly dose-dense regimen vs the standard regimen, as per randomization Addition of bevacizumab to chemotherapy, as per investigator decision Late debulking surgery after chemotherapy in the case of favorable response to chemotherapy, as per investigator decision Maintenance treatment with bevacizumab with/without PARP inhibitor, or surveillance, as per investigator decision
Incremental cost-effectiveness ratio | from date of randomization until end of study, for a period of 5 years
  To assess the cost-effectiveness evaluations of the experimental treatment (medico-economic evaluation) in the French context Salvage weekly dose-dense regimen vs the standard 3-weekly regimen, as per randomization Addition of bevacizumab to chemotherapy, as per investigator decision Late debulking surgery after chemotherapy in the case of favorable response to chemotherapy, as per investigator decision Maintenance treatment with bevacizumab with/without PARP inhibitor, or surveillance, as per investigator decision
Estimate the net financial impact over 5 years | from date of randomization until end of study, for a period of 5 years
  A budget impact analysis (BIA) to estimate the financial impact for French Health Insurance of the generalization in the French context of the strategy based on the experimental treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit YOU, Principal Investigator — HCL - Centre Hospitalier Lyon Sud
Locations (72):
- France (50):
  - ICO Paul Papin, Angers
  - CH d'Avignon, Avignon
  - Sainte-Catherine Institut du Cancer Avignon-Provence, Avignon
  - Hôpital de la Côte Basque, Bayonne
  - CHRU Besançon - Hôpital Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - CHU de BREST - Hôpital Cavale Blanche, Brest
  - Centre François Baclesse, Caen
  - Centre d'Oncologie et de Radiothérapie 37 (ROC37), Chambray-lès-Tours
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - CHU de Dijon, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Hôpital André Mignot, Le Chesnay
  - CHRU de Lille, Lille
  - Centre Oscar Lambret, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Hôpital de la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - Hôpital de la Timone, Marseille
  - CHRU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - ICM Val d'Aurelle, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - Hôpital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut de Cancérologie du Gard - CHU de Nîmes, Nîmes
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Hôpital Cochin, Paris
  - Hôpital Européen George Pompidou, Paris
  - Institut Curie, Paris
  - Centre Hospitalier Général de Pau, Pau
  - HCL - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital de Poissy-Saint-Germain-en-Laye, Poissy
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Hôpital Privé de la Loire, Saint-Etienne
  - Institut de Cancérologie de l'Ouest - ICO, Saint-Herblain
  - CHU Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - CHU Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpitaux du Léman - site Thonon-les-Bains, Thonon-les-Bains
  - Oncopole Claudius Régaud - IUCT Oncopole, Toulouse
  - Clinique Pasteur, Toulouse
  - Centre Hospitalier de Valence, Valence
  - Gustave Roussy, Villejuif
- Italy (6):
  - Azienda Ospedaliero-Universitaria Ss.Antonio E Biagio E C.Arrigo Alessandria, Alessandria
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS Istituto Di Ricerca E Di Cura A Carattere Scientifico, Bologna
  - Careggi University Hospital, Florence
  - Alessandro Manzoni Hospital, Lecco
  - Istituto Europeo Di Oncologia S.r.l., Milan
  - Azienda Ulss 3 Serenissima, Venice
- Japan (16):
  - The University of Tokyo Hospital, Bunkyō City
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Medical University International Medical Center, Hidaka
  - Hirosaki University Hospital, Hirosaki
  - The Jikei University Kashiwa Hospital, Kashiwa
  - St. Marianna University Hospital, Kawasaki
  - Dokkyo Medical University Saitama Medical Center, Koshigaya
  - Kurume University Hospital, Kurume
  - Nagoya University Hospital, Nagoya
  - Kindai University Hospital, Sayama
  - Tohoku University Hospital, Sendai
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - The Cancer Institute Hospital Of JFCR, Tokyo
  - The Jikei University Daisan Hospital, Tokyo
  - The Jikei University Hospital, Tokyo
  - The Jikei University Katsushika Medical Center, Tokyo

REFERENCES:
- [Derived] Chator C, Yanaihara N, Chabaud S, Parma GM, Dima AL, Clamp A, Ferron G, Kroep JR, Leary A, Cibula D, Fiteni F, Bruchim I, Serrier H, Carroll S, Belmont AS, Peron J, You B. SALVOVAR: a pragmatic randomized phase III trial comparing the SALVage weekly dose-dense regimen to the standard 3-weekly regimen in patients with poor prognostic OVARian cancers. Ther Adv Med Oncol. 2025 Dec 23;17:17588359251396777. doi: 10.1177/17588359251396777. eCollection 2025. PMID 41466844